CLINICAL TRIAL: NCT00774826
Title: Phase III Multicentric IIL Study, Three Randomized Arms (R-CVP vs R-CHOP vs R-FM),for Treatment of Patients With Stage II-IV Follicular Lymphoma
Brief Title: Multicentric Study, Three Randomized Arms (R-CVP vs R-CHOP vs R-FM),for Patients With Stage II-IV Follicular Lymphoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fondazione Italiana Linfomi - ETS (Other)
Responsible Party: MASSIMO FEDERICO, AZIENDA OSPEDALIERA POLICLINICO - MODENA (MO)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIL-FOLL05; Eudract Number 2005-005406-24
Record Dates: First submitted 2008-10-14; First posted 2008-10-17 (Estimated); Last update posted 2011-02-15 (Estimated); Status verified 2011-02

CONDITIONS: Follicular Lymphoma
Keywords: Follicular lymphoma; Rituximab
MeSH Terms: conditions — Lymphoma, Follicular | interventions — R-CHOP protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): R-CVP x 3; Restaging if> RP then R-CVP x 5
  Interventions: Drug: R-CVP
- 2 (Experimental): R-CHOP x 3; Restaging if > RP then R-CHOP x 3 plus 2 Rituximab
  Interventions: Drug: R-CHOP
- 3 (Experimental): R-FM x 3; Restaging if > RP then R-FM x 3 plus 2 Rituximab
  Interventions: Drug: R-FM

INTERVENTIONS:
Drug: R-CVP — Rituximab: 375 mg/mq day 1 Ciclofosfamide: 750 mg/mq day 1, Vincristina: 1,4 mg/mq day 1 Prednisone: 40 mg/mq day 1-5,
  Arms: 1
Drug: R-CHOP — Rituximab: 375 mg/mq day 1 Ciclofosfamide: 750 mg/mq day 1 Doxorubicina: 50 mg/mq day 1 Vincristina: 1.4 mg/mq day 1 Prednisone: 100 mg/mq day 1-5
  Arms: 2
Drug: R-FM — Rituximab: 375 mg/mq day 1, Fludarabina: 25 mg/mq day 1-3, Mitoxantrone: 10 mg/mq day 1,
  Arms: 3

SUMMARY:
The purpose of this study is to define an improvement and theassessment of the Time to Treatment Failure in patients randomized in three different arms:

R-CVP vs R-CHOP vs R-FM.

DETAILED DESCRIPTION:
Assessment of Overall Survival (OS)in patients treated with R-CVP, R-CHOP and R-FM. -Assessment of Progression Free Survival (PFS)in patients treated with R-CVP, R-CHOP - Assessment of Duration of Response (DR)in patients treated with R-CVP, R-CHOP and R-FM. - Assessment of Response Rate(RR) in patients treated with R-CVP, R-CHOP and R-FM. - Assessment of molecular Response Rate in patients treated with R-CVP, R-CHOP and R-FM. - Assessment of toxicity of R-CVP, R-CHOP, R-FM treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Histological DIAGNOSIS of B cell follicular lymphoma
2. ECOG performance status 0-2
3. Age range 18-75
4. Ann Arbor Stage: II-IV
5. Assessment of pathology with diagnostics biopsy
6. Presence of one of these criteria:

   * B Sistemic symptoms B
   * Extranodale pathology
   * Cytopenia
   * Splenomegaly
   * Leukemia
   * Serous effusion
   * Ves > 20 mm/h
   * Ldh > normal value
   * Nodale or extranodal mass > 7 cm
   * 3 or more nodal sites > 3 cm
   * Adenopatic syndrome
7. LVEF > 50%
8. Normal hepatic (bilirubin < 1.5 mg/dl) and renal functionality (creatinin < 2 mg/dl). If there is a lymphoma it's allow values of bilirubin > 1.5 mg/dl and of creatinin > 2mg/dl
9. No previous treatment for follicolar lymphoma unless RT-IF
10. Lifetime > 6 mounth
11. Absence of HbsAg, HCV e HIV
12. Negative Coombs Test
13. Negative pregnant test
14. Cotracceptive method during the treatment and the follow three months
15. Formal written consent
16. Ability to follow the patients after the treatment for follow up

Exclusion Criteria:

1. Histological Diagnosis of all type of lymphoma unless Follicularlymphoma, CD20 lymphoma, stage IIIb of follicular lymphoma and high degree lymphoma
2. Stage I of Ann Arbor scale
3. Central Nervous system involvement
4. HIV, HBV OR HCV Positivity
5. Cardiac Pathology
6. Positive Coombs Test
7. Previous chemotherapeutic treatment
8. Hypersensitivity to antibodyes or other murine proteins
9. Previous cancer pathology unless in situ cervix and epithelial carcinomas
10. Other type of infections
11. Pregnant and nursing woman

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 534 (Actual)
Dates: Start 2005-12; Primary Completion 2010-09 (Actual); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Assessment of the Time to Treatment Failure (TTF)in patients treated with R-CVP, R-CHOP and R-FM. | 2 years

SECONDARY OUTCOMES:
Assessment of Overall Survival (OS)in patients treated with R-CVP, R-CHOP and R-FM. - | 3 years
Assessment of Progression Free Survival (PFS)in patients treated with R-CVP, R-CHOP | 2 years
Assessment of Duration of Response (DR)in patients treated with R-CVP, R-CHOP and R-FM. | 2 years
Assessment of Response Rate(RR) in patients treated with R-CVP, R-CHOP and R-FM. | 2 years
Assessment of molecular Response Rate in patients treated with R-CVP, R-CHOP and R-FM. | 2 years
Assessment of toxicity of R-CVP, R-CHOP, R-FM treatments. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Federico, PhD, Principal Investigator — Azienda Ospedaliero-Universitaria di Modena
Locations (82):
- Italy (82):
  - Azienda Ospedaliera S. Maria, Terni, Terni
  - Ente ecclesiastico Ospedale generale regionale Miulli, Acquaviva Delle Fonti (BA)
  - Az.Ospedaliera SS.Antonio, Biagio e Cesare Arrigo-U.O.A.Ematologia, Alessandria
  - Presidio Ospedaliero C.Massaia di Asti, Asti
  - Istituto Nazionale Tumori, Aviano
  - IRCCS Istituto tumori Giovanni Paolo II, Bari
  - Divisione Medicina B Ospedale degli Infermi, Biella
  - Policlinico Sant'Orsola - Istituto di Ematologia e Oncologia medica L.e A. Seragnoli, Bologna
  - Ospedale di Bolzano Divisione di Ematologia e Centro Trapianti di Midollo Osseo, Bolzano
  - A.O.Spedali civili di Brescia, Brescia
  - Presidio Ospedaliero A.Perrino, Brindisi
  - Ospedale Businco, Divisione di Ematologia, Cagliari
  - Ospedale Civile, Camposanpiero (PD)
  - Istituto per la ricerca e la cura del cancro, Candiolo (TO)
  - A.O. dell'Annunziata Unita' Operativa di Ematologia, Carpi (MO)
  - Ospedale Ramazzini Day Hospital Oncologico, Carpi (Mo)
  - Ospedale Garibaldi-Nesima, Catania
  - Universita' degli studi di Catania, Catania
  - A.O. Pugliese A. Ciaccio, Catanzaro
  - A.O.Pugliese Ciaccio Diviisone di Ematologia, Catanzaro
  - Ospedale civico di Chivasso, Chivasso (TO)
  - Ospedale di Ciriè U.O.N.A. Oncologia servizio di Ematologia, Ciriè (TO)
  - Ospedale civile Divisione di Ematologia, Civitanova Marche (MC)
  - Ospedale San Sebastiano, Correggio (RE)
  - Presidio Ospedaliero Annunziata, Cosenza
  - Azienda istituti ospedalieri di Cremona, Cremona
  - Policlinico Careggi, cattedra e diviisone di Ematologia, Florence
  - E.O.Ospedali Galliera U.O.Ematologia, Genova
  - Ospedale San Martino - Divisione di Ematologia, Genova
  - Ospedale Felettino reparto di Oncologia, La Spezia
  - Ospedale Vito Fazzi, Lecce
  - Ospedale A.Manzoni Oncologia medica, Lecco
  - Ospedale Madonna delle grazie U.O. Ematologia, Matera
  - Azienda Ospedaliera Papardo, Messina
  - Policlinico universitario U.O. Ematologia, Messina
  - Azienda Ospedaliera Fatebenefratelli e Oftalmico, Milan
  - IRCCS San Raffaele Unità di Chemioterapia, Milan
  - Osp. San Carlo Borromeo Divisione di Oncologia Medica, Milan
  - Ospedale Maggiore IRCCS-Dipartimento di Ematologia, Milan
  - Ospedale Niguarda CA' Granda, Milan
  - Ospedale San Paolo U.O. Oncologia Medica, Milan
  - Policlinico di Modena - Università degli studi, Modena
  - Ospedale S. Gerardo Divisione di ematologia, Monza (MI)
  - AORN Cardarelli U.O.Ematologia, Napoli
  - Ospedale P.F.Calvi dipartimento id Oncologia ed Ematologia, Noale
  - Presidio Ospedaliero Umberto I Medicina ed Onco-Ematologia, Nocera Inferiore
  - A.O. Maggiore della Carità S.C.D.U. Ematologia, Novara
  - A.O. di Padova Divisione di Oncologia Medica, Padua
  - Casa di cura La Maddalena Unita' di Ematologia, Palermo
  - Policlinico P.Giaccone, Palermo
  - Universita' degli studi di Parma, Parma
  - Policlinico San Matteo - Medicina generale, Pavia
  - Policlinico San Matteo, Pavia
  - Policlinico Monteluce Divisione di Ematologia, Perugia
  - Ospedale Santo Spirito Dipartimento di Ematologia, Pescara
  - Ospedale Santo Spirito-Dipartimento di Oncologia, Pescara
  - Ospedale Civile, Sezione di Ematologia, Piacenza
  - Ospedale S. Chiara Azienda ospedaliera pisana, Pisa
  - Presidio Ospedali riuniti "Bianchi, Melacrino, Morelli" Divisione di ematologia, Reggio Calabria
  - Azienda ospedaliera Arcispedale S.Maria Nuova, Reggio Emilia
  - Ospedale Oncologico regionale CROB, Rionero in Vulture (PZ)
  - A.O.S.Andrea Reparto di Ematologia e Immunoematologia, Roma
  - Azienda Policlinico Umberto I - La Sapienza, Roma
  - Istituto Regina Elena, Roma
  - Ospedale San Giacomo U.O. Ematologia, Roma
  - Policlinico A. Gemelli Università Cattolica del Sacro Cuore, Roma
  - Policlinico Universitario Campus biomedico, Roma
  - Policlinico Universitario Tor Vergata, Roma
  - Universita' La Sapienza, Roma
  - P.O. Roncilgione U.O. Ematologia, Ronciglione (VT)
  - Istituto clinco Humanitas, Rozzano (MI)
  - IRCCS Casa Sollievo della Sofferenza, San Giovanni Rotondo (FG)
  - Istituto di Ematologia Università degli studi di Sassari, Sassari
  - Ospedale civile DH oncologico, Sassuolo (MO)
  - Ospedale San Paolo, Savona
  - A.O. della Valtellina e della Valchiavenna Presidio Ospedaliero di Sondalo, Sondalo
  - Ospedale S. Maria Clinica Medica Servizio Oncologico, Terni
  - A.O.San Giovanni Battista, Torino
  - A.O.Cardinale Panico Ematologia e centro trapianti, Tricase (LE)
  - Azienda Ospedaliera Ospedali riuniti di Trieste, Trieste
  - Ospedale di circolo e Fondazione Macchi, Varese
  - O.C.SS. Giovanni e Paolo - U.O. Ematologia, Venezia

REFERENCES:
- [Derived] Luminari S, Ferrari A, Manni M, Dondi A, Chiarenza A, Merli F, Rusconi C, Tarantino V, Tucci A, Vitolo U, Kovalchuk S, Angelucci E, Pulsoni A, Arcaini L, Angrilli F, Gaidano G, Stelitano C, Bertoldero G, Cascavilla N, Salvi F, Ferreri AJM, Vallisa D, Marcheselli L, Federico M. Long-Term Results of the FOLL05 Trial Comparing R-CVP Versus R-CHOP Versus R-FM for the Initial Treatment of Patients With Advanced-Stage Symptomatic Follicular Lymphoma. J Clin Oncol. 2018 Mar 1;36(7):689-696. doi: 10.1200/JCO.2017.74.1652. Epub 2017 Nov 2. PMID 29095677
- [Derived] Rossi D, Bruscaggin A, La Cava P, Galimberti S, Ciabatti E, Luminari S, Rigacci L, Tucci A, Pulsoni A, Bertoldero G, Vallisa D, Rusconi C, Spina M, Arcaini L, Angrilli F, Stelitano C, Merli F, Gaidano G, Federico M, Palumbo GA. The genotype of MLH1 identifies a subgroup of follicular lymphoma patients who do not benefit from doxorubicin: FIL-FOLL study. Haematologica. 2015 Apr;100(4):517-24. doi: 10.3324/haematol.2014.108183. Epub 2015 Jan 16. PMID 25596266